CLINICAL TRIAL: NCT00336154
Title: Randomised Double Blind Crossover Placebo Controlled Study to Evaluate the Efficacy of Tetracycline in Epidermolysis Bullosa
Brief Title: Study to Evaluate the Efficacy of Tetracycline in Epidermolysis Bullosa
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Sponsor: Rambam Health Care Campus (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 2140CTIL
Record Dates: First submitted 2006-06-12; First posted 2006-06-13 (Estimated); Last update posted 2020-10-28 (Actual); Status verified 2020-10

CONDITIONS: Epidermolysis Bullosa
MeSH Terms: conditions — Epidermolysis Bullosa | interventions — Tetracycline

INTERVENTIONS:
Drug: tetracyclin

SUMMARY:
Epidermolysis Bullosa(EB) is an inherited bullous disease. Tetracycline is believed to have anti inflammatory properties. 20 patients with EB older than 13 years will be treated for 4 months with tetracycline or placebo. After one month of wash out they will be treated for additional 4 m with placebo or tetracycline. The patients will be examined each month to estimate bulla formation,rate of healing .

DETAILED DESCRIPTION:
Epidermolysis Bullosa(EB) is an inherited bullous disease. Tetracycline is believed to have anti inflammatory properties. 20 patients with EB older than 13 years will be treated for 4 months with tetracycline or placebo. After one month of wash out they will be treated for additional 4 m with placebo or tetracycline. The patients will be examined each month to estimate bulla formation,rate of healing .

ELIGIBILITY:
Inclusion Criteria:

* diagnosed as epidermolysis bullosa
* not pregnant
* active disease
* more than 5 bulla-

Exclusion Criteria:

* age less than 13
* known sensitivity to tetracyclin
* abnormal liver and kidney tests.

Ages: 13 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Primary Completion 2006-06 (Estimated)

PRIMARY OUTCOMES:
no of blisters